CLINICAL TRIAL: NCT01246947
Title: A Prospective Randomized Trial of Tricuspid Annuloplasty for Moderate Tricuspid Regurgitation Associated With Mitral Operation
Brief Title: Tricuspid Annuloplasty for Moderate Tricuspid Regurgitation Associated With Miral Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00044723
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2017-06

CONDITIONS: Cardiac Surgery; Tricuspid Valve Regurgitation
Keywords: Moderate Tricuspid Valve Regurgitation; Tricuspid Valve Repair; Mitral Value Surgery
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitral surgery alone (Active Comparator): Mitral valve surgery randomization for no repair of the moderate tricuspid regurgitation
  Interventions: Other: Mitral surgery alone
- Mitral surgery w/Tricuspid valve repair (Active Comparator): Mitral valve surgery with randomization to repair the moderate tricuspid regurgitation
  Interventions: Procedure: Tricuspid valve repair

INTERVENTIONS:
Procedure: Tricuspid valve repair — Randomized to receive Tricuspid valve repair using a rigid 3-dimensional annuloplasty ring using standard techniques, during Mitral surgery.
  Other Names: Tricuspid valve annuloplasty
  Arms: Mitral surgery w/Tricuspid valve repair
Other: Mitral surgery alone — Randomized to Mitral surgery alone
  Arms: Mitral surgery alone

SUMMARY:
The mitral valve is the inflow valve into the main pumping chamber of the heart. It can become leaky or narrow, and cause blood to back up into the blood vessels of the lungs. When patients get symptoms from a leaky or narrow mitral valve, surgery is recommended to either fix or replace the valve. Many patients with mitral valve disease also develop a leaky tricuspid valve - the tricuspid valve is the inflow valve to the right side of the heart (the right heart pumps blood across the lungs). The amount of leakiness of the tricuspid valve is determined by an ultrasound test, and the amount of leakiness is graded as: none, mild, moderate, or severe. When a heart surgeon operates on a patient with a diseased mitral valve, he or she will fix the tricuspid valve if the tricuspid leakage is severe. This involves sewing a cloth-covered ring around the valve and narrowing it. If the tricuspid valve leakage is only mild (or absent), the surgeon will leave the tricuspid valve alone at the time of mitral valve surgery. If the tricuspid valve has moderate leakage surgeons are uncertain about what to do. In a recent review of thousands of patients across the nation having mitral valve surgery with moderately leaky tricuspid valves, 35 % of patients had tricuspid valve repair. Since the investigators don't know what the best approach is: to leave the moderately leaky tricuspid valve alone or to fix it with a cloth-covered ring, the investigators propose a study to determine which approach is best. Patients having mitral valve surgery with a moderately leaky tricuspid valve will be randomized to either 1. have a tricuspid valve repair or 2. to not have a tricuspid valve repair. The investigators will carefully follow these patients for two years and see if heart function is better among those who got their valve fixed.

DETAILED DESCRIPTION:
Study Design:

This is a single-center prospective, randomized controlled clinical trial.

Enroll/Randomize: mitral operation alone, or mitral operation with tricuspid valve repair. Randomization will occur before operation.

Operation: The surgeon will perform mitral surgery and only those patients randomized to tricuspid valve repair will perform tricuspid valve repair using a rigid 3-dimensional annuloplasty ring using standard techniques.

ELIGIBILITY:
Inclusion Criteria:

1. All patients 18-65 + older years undergoing mitral valve surgery.
2. Presence of moderate or mild-moderate tricuspid regurgitation as read on any echocardiographic study performed within 6 months prior to operation. Assessment if tricuspid regurgitation will be performed using an integrative method.
3. All patients referred for mitral valve surgery.
4. Able to understand the consent and able to sign informal consent.

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patient with structural/ organic tricuspid valve disease.
3. Refusal/ Inability to sign informal consent form.
4. Pregnant women.
5. Tricuspid valve endocarditis.
6. Requirement for concomitant cardiac surgery (other than atrial fibrillation correction surgery, closure of PFO (Patent Foramen Ovale) or ASD (Atrial Septal Defect), or coronary artery bypass surgery).
7. Cardiogenic shock at the time of randomization.
8. ST segment elevation myocardial infarction requiring Intervention within 7 days prior to randomization.
9. Evidence of cirrhosis or hepatic synthetic failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The degree of tricuspid regurgitation at 12 months after surgery | 12 months
  Standard transthoracic echocardiographic assessment of the degree of tricuspid regurgitation will be performed as described in "Recommendations for evaluation of the severity of native valvular regurgitation with two-dimensional and Doppler echocardiography" (Zoghbi et al, J Am Soc Echocardiography 2003; 16:777-802).
  An integrative approach will be used, and patients will be categorized as having one of:
  1. none/trivial
  2. mild
  3. moderate
  4. severe Tricuspid regurgitation.

SECONDARY OUTCOMES:
NYHA heart failure functional status | 12 Months
  New York Heart Association Classification (NYHA)Class Class I (Asymptomatic)No limitation of ordinary physical activity. Class II (Mild)Slight limitation. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III (Moderate)Marked limitation. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV (Severe)Unable to carry out any physical activity without discomfort.
NYHA heart failure functional status | 24 Months
  New York Heart Association Classification (NYHA)Class Class I (Asymptomatic)No limitation of ordinary physical activity. Class II (Mild)Slight limitation. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  Class III (Moderate)Marked limitation. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV (Severe)Unable to carry out any physical activity without discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: James S Gammie, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Result] Zoghbi WA, Enriquez-Sarano M, Foster E, Grayburn PA, Kraft CD, Levine RA, Nihoyannopoulos P, Otto CM, Quinones MA, Rakowski H, Stewart WJ, Waggoner A, Weissman NJ; American Society of Echocardiography. Recommendations for evaluation of the severity of native valvular regurgitation with two-dimensional and Doppler echocardiography. J Am Soc Echocardiogr. 2003 Jul;16(7):777-802. doi: 10.1016/S0894-7317(03)00335-3. No abstract available. PMID 12835667